CLINICAL TRIAL: NCT03244280
Title: A Study of the Systemic Absorption of Once Daily MOB015B When Applied for 28 Days in Subjects With Moderate to Severe Onychomycosis of the Toenails.
Brief Title: A Study of the Systemic Absorption of MOB015B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MOB015B-VIII
Record Dates: First submitted 2017-08-01; First posted 2017-08-09 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MOB015B (Other)
  Interventions: Drug: MOB015B

INTERVENTIONS:
Drug: MOB015B — Topical formulation

SUMMARY:
A Study of the Systemic Absorption of Once Daily MOB015B when Applied for 28 Days in Subjects with Moderate to Severe Onychomycosis of the Toenails.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand the study procedures and agree to participate by providing written informed consent. Subject must be willing to authorize use and disclosure of protected health information collected for the study.
2. Male or female subjects 12 to 70 years of age (inclusive), at the time of consent.
3. Subject has a body mass index (BMI) from ≥ 18.5 to ≤ 35.0 (kg/m2), at the screening visit.
4. Females of childbearing potential must be using contraception during the study which can include abstinence or hormonal contraceptives. All women of childbearing potential must be willing to complete a urine pregnancy test on Days 1, 14, and 28.
5. Subjects must present with a clinical diagnosis of moderate to severe subungal onychomycosis with at least 50% involvement of both great toenails. In addition, 4 other toenails must be affected.
6. Subjects must have a positive KOH microscopy for at least 1 great toenail at the screening visit.
7. Subjects must be willing to complete clinical laboratory testing.
8. Subjects must be willing to undergo alcohol and drug (e.g., benzodiazepines, cocaine, opioids, cannabinoids, and barbiturates) tests at the Day 1 visit.
9. Subjects must be willing to remain at the study site for approximately 11 hours and undergo multiple blood draws on Day 1 and 28.
10. Subjects must be able to reach their toes to apply study drug or have a caregiver willing to help apply the study drug on a daily basis as directed.

Exclusion Criteria:

1. Female subjects who are pregnant, nursing/breastfeeding, or plan to become pregnant within the study period.
2. Subjects with chronic or active liver disease, renal impairment, cutaneous or systematic lupus erythematosus, or any other disease or medical condition that in the opinion of the investigator would interfere with the study or place the subject at undue risk.
3. Subject with hypersensitivity to terbinafine or the vehicle excipients.
4. Subjects who have been treated with systematic formulations of terbinafine in the 12 months prior to the Day 1 visit.
5. Subjects who have been treated with topical formulations of terbinafine in the 6 months prior to the day 1 visit.
6. Subjects who take or have taken systematic medication that may interfere with the study or place the subject at undue risk in the 30 days before the day 1 visit (e.g., rifampin, cimetidine, phenobarbital, phenytoin, carbamazepine, terfenadine or digoxin).
7. Subjects who take or have taken systemic medication in the 30 days before the Day 1 visit that interferes with the terbinafine plasma assay.
8. Subjects who have consumed grapefruit products during the 30 days prior to the Day 1 visit.
9. Subjects who are not willing to refrain from caffeinated beverage consumption on Day 1 and 28.
10. Subjects with a current history of consumption of more than three alcoholic drinks per day or consumption of alcohol within 48 hours prior to Day 1 visit (one drink is equal to one unit of alcohol, one glass of wine, half pint of beer or one ounce of spirits).
11. Subjects with an ongoing or recent history of treatment for substance abuse.
12. Subjects who have participated in a study of an investigational drug 60 days prior to the Day 1 visit.
13. Subjects with a history of multiple syncopal episodes.
14. Subjects with positive tests for drugs or alcohol at Day 1 visit.
15. Subjects who are unable to comply with study requirements.
16. Subjects who are not willing to abstain from all toenail treatments such as toenail polish, pedicures and/or foot soaks (including nail clipping or debridement), for 3 days prior to Day 1 visit and during the study.
17. Donation of blood (one unit or 350 mL) within 90 days prior to Day 1 visit.

    -

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-16 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
To measure the Cmax | 28 days
  To measure the Cmax after 1 day and 28 days
To measure the Tmax | 28 days
  To measure Tmax after 1 day and 28 days
to measure AUC0-t | 28 days
  To measure AUC0-t after 1 day and 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tavakkol A, DuBois JC, Gupta AK. Systemic absorption and safety of topical terbinafine hydrochloride 10% solution (MOB015B): a phase 1 maximal usage trial in patients with moderate-to-severe onychomycosis. Antimicrob Agents Chemother. 2024 Oct 8;68(10):e0068224. doi: 10.1128/aac.00682-24. Epub 2024 Aug 19. PMID 39158295